CLINICAL TRIAL: NCT04661215
Title: Pyloric Sphincter Abnormalities in Patients With Gastroparesis Symptoms
Acronym: PSAGS
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Massachusetts General Hospital (Other); Temple University (Other); University of Louisville (Other); Wake Forest University (Other); Texas Tech University Health Sciences Center, El Paso (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 12 DK PSAGS; U24DK074008 (NIH); U01DK073974 (NIH); U01DK074007 (NIH); U01DK074035 (NIH); U01DK073975 (NIH); U01DK112193 (NIH); U01DK073983 (NIH)
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gastroparesis; Idiopathic Gastric Motility Disorder; Diabetic Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Symptoms of gastroparesis: Participants with symptoms of gastroparesis with minimum Gastroparesis Cardinal Symptom Index (GCSI) score of 2.0
- Control participants: Participants undergoing endoscopy for evaluation but without gastroparesis symptoms or gastroesophageal reflux symptoms. Score 1.0 or less (≤ 1 ) on the GCSI of Patient Assessment of Upper Gastrointestinal Symptom Severity Index (PAGI-SYM) questionnaire

SUMMARY:
The overall objective of this study is to determine if there are pyloric sphincter abnormalities in patients with gastroparesis symptoms and determine how prevalent these abnormalities are using tests to assess the pyloric sphincter - endoluminal functional luminal imaging probe (Endoflip™), water load satiety testing (WLST), and high-resolution cutaneous electrogastrography (HR-EGG) using Gastric Alimetry™ System.

DETAILED DESCRIPTION:
Study Description: This is a multi-center, prospective, observational study to assess pyloric sphincter abnormalities in patients with symptoms of gastroparesis (both delayed and normal gastric emptying) and control participants without symptoms of gastroparesis using the commercially available, FDA approved endoluminal functional luminal imaging probe (Endoflip™) catheter, which measures diameter, cross-sectional area, pressure, compliance, and distensibility of gastrointestinal sphincter muscles.

This study will assess lower esophageal and pyloric sphincter diameter, CSA, pressure, distensibility, and compliance in patients with symptoms of gastroparesis and delayed gastric emptying, patients with symptoms of gastroparesis but with normal gastric emptying, and normal control participants. The protocol will also include a water load satiety test and use Gastric Alimetry™ System that assesses gastric myoelectrical activity in symptomatic participants but not control participants.

ELIGIBILITY:
Inclusion Criteria FOR SYMPTOMATIC PARTICIPANTS:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18-85
4. Symptoms of gastroparesis, either diabetic or idiopathic etiology
5. Symptoms of gastroparesis with minimum Gastroparesis Cardinal Symptom Index (GCSI) score of 2.0
6. Individual will have had a prior 4-hour gastric emptying scintigraphy test performed for clinical evaluation within the last 6 months. This gastric emptying test would be done for clinical evaluation and is not part of the research study. From these participants with gastroparesis symptoms, we will include those with delayed gastric emptying as well as those with normal gastric emptying.
7. Participant must not initiate any new treatments until completion of the study procedures.
8. Willingness to:

   1. Stop histamine 2 antagonists, prokinetics (e.g., metoclopramide, erythromycin, domperidone, prucalopride), narcotics, anticholinergics, constipation medications (over the counter laxatives, isotonic polyethylene glycol (PEG) electrolyte preparations (e.g. MiraLax), prescription laxatives (e.g. lubiprostone), proton pump inhibitors, cannabinoids, and cannabidiol (CBD) for 3 days prior to each visit;
   2. Abstain from food and water after midnight (at least for 8 hours) before the start of each visit until after the visit.

INCLUSION CRITERIA FOR CONTROL PARTICIPANTS

1. Provision of signed and dated informed consent form
2. Male or female, aged 18 or older
3. Undergoing an upper endoscopy for their clinical evaluation of diarrhea, GI bleed, or iron-deficiency anemia, or evaluation for bariatric surgery.
4. Do not have upper GI symptoms greater than 1 as assessed by the Gastroparesis Cardinal Symptom Index (GCSI) of PAGI-SYM questionnaire.

EXCLUSION CRITERIA:

1. Prior gut lumen surgery on the esophagus or the stomach, including Nissen fundoplication.
2. Prior surgery on the pylorus (G-POEM, surgical pyloroplasty, surgical pyloromyotomy)
3. Known history of achalasia or esophageal stricture
4. Known history of physiological or mechanical GI obstruction
5. Abnormalities seen on a prior upper endoscopy placing patient at increased risk:

   * Ulcer of the esophagus, stomach, or duodenum
   * Esophageal varices
6. Individuals at risk for prolonging the endoscopy procedure: severe chronic pulmonary disease, severe food retention in the stomach on endoscopy.
7. Presence of significant gastric or duodenal pathology that could be expected to cause dysmotility (e.g. significant inflammation, infiltrate disorders etc)
8. Individuals with a history of other chronic disease potentially causative of gastrointestinal symptom
9. Acute or chronic renal insufficiency
10. Current eating disorders
11. Females who are pregnant. A urine pregnancy test is routinely obtained on all females immediately prior to endoscopic procedures.
12. Individuals with contraindications for endoscopy, including bleeding abnormalities
13. Allergy to eggs preventing sedation with propofol and/or gastric emptying test
14. Significant dysphagia
15. Prior inflammatory bowel disease, Crohn's
16. History of any esophageal/gastric/pyloric injection of botulinum toxin
17. Patients on daily opioid use or >3 day/week use
18. Use of glucagon-like peptide 1 (GLP1) receptor agonists or Sodium-Glucose Transport Protein 2 (SGLT2); Gastric inhibitory polypeptide (GIP)- glucagon-like peptide (GLP) combo

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be 150 adult men and women aged 18-85 years, located in the United States, 100 will have symptoms of gastroparesis, and 50 participants in the control group will be patients undergoing upper endoscopy for clinical evaluation of diarrhea, gastrointestinal (GI) bleed, or iron-deficiency anemia, or evaluation for bariatric surgery who do not have upper GI symptoms greater than 1 as assessed by the Gastroparesis Cardinal Symptom Index (GCSI) . Control group participants will not have Gastric Alimetry testing or water load satiety testing.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Distensibility of the pylorus | Baseline
  Distensibility of the pylorus will be calculated as the median of three measurements (not three different inflations) of distensibility (mm2/mmHg) of the pylorus pressure using the Endoflip balloon catheter at 50 mL volume

SECONDARY OUTCOMES:
Opening diameter (mm) of the pylorus when 40 mL volume is introduced into the EF325N Endoflip™ measurement catheter. | Baseline
  diameter (mm) of the pylorus
Opening diameter (mm) of the pylorus when 50 mL volume is introduced into the EF325N Endoflip™ measurement catheter. | Baseline
  diameter (mm) of the pylorus
Cross Sectional Area(mm2) of the pylorus with 40 mL balloon volume | Baseline
  Cross Sectional Area (mm2) of the pylorus
Cross Sectional Area(mm2) of the pylorus with 50 mL balloon volume | Baseline
  Cross Sectional Area (mm2) of the pylorus
Compliance (mm3/mmHg) of the pylorus with 40 mL balloon volume | Baseline
  Compliance (mm3/mmHg) of the pylorus
Compliance (mm3/mmHg) of the pylorus with 50 mL balloon volume | Baseline
  Compliance (mm3/mmHg) of the pylorus
Pressure (mmHg) of the pyloric sphincter | Baseline
  Pressure (mmHg) of the pyloric sphincter

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Pasricha, MD, Study Chair — Mayo Clinic; Henry Parkman, MD, Study Chair — Temple University
Locations (6):
- United States (6):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of Louisville, Louisville, Kentucky
  - Massachusetts General, Boston, Massachusetts
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - Texas Tech University Health Science Center (TTUHSC), El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Public use complete database will be submitted to the NIDDK Data Repository
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: By the end of the funding period
Access Criteria: Application through National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository; Institutional Review Board (IRB) approval
URL: https://repository.niddk.nih.gov/home

REFERENCES:
- [Background] Fisher R, Cohen S. Physiological characteristics of the human pyloric sphincter. Gastroenterology. 1973 Jan;64(1):67-75. No abstract available. PMID 4683856
- [Background] Parkman HP, Hasler WL, Fisher RS; American Gastroenterological Association. American Gastroenterological Association technical review on the diagnosis and treatment of gastroparesis. Gastroenterology. 2004 Nov;127(5):1592-622. doi: 10.1053/j.gastro.2004.09.055. PMID 15521026
- [Background] Desipio J, Friedenberg FK, Korimilli A, Richter JE, Parkman HP, Fisher RS. High-resolution solid-state manometry of the antropyloroduodenal region. Neurogastroenterol Motil. 2007 Mar;19(3):188-95. doi: 10.1111/j.1365-2982.2006.00866.x. PMID 17300288
- [Background] Mearin F, Camilleri M, Malagelada JR. Pyloric dysfunction in diabetics with recurrent nausea and vomiting. Gastroenterology. 1986 Jun;90(6):1919-25. doi: 10.1016/0016-5085(86)90262-3. PMID 3699409